CLINICAL TRIAL: NCT01969721
Title: Randomized, Double-blind, Double-dummy, Active-controlled, 4 Period Complete Cross-over Study to Compare the Effect on Lung Function of 6 Weeks Once Daily Treatment With Orally Inhaled Tiotropium+Olodaterol Fixed Dose Combination Delivered by the Respimat® Inhaler vs. 6 Weeks Twice Daily Treatment With Fluticasone Propionate+Salmeterol Fixed Dose Combination Delivered by the Accuhaler® in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Characterization of Lung Function Profile of Inhaled Tiotropium + Olodaterol Fixed Dose Combination Compared to Fluticasone Propionate + Salmeterol Fixed Dose Combination in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.11; 2013-000808-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate; Tiotropium Bromide; olodaterol

ARMS (4):
- T+O FDC dosage 1 (Experimental): Low dose
  Interventions: Drug: olodaterol; Drug: placebo; Drug: tiotropium
- T+O FDC dosage 2 (Experimental): High dose
  Interventions: Drug: placebo; Drug: tiotropium; Drug: olodaterol
- ICS/LABA FDC Dosage 1 (Active Comparator): Low dose
  Interventions: Drug: fluticasone propionate; Drug: salmeterol; Drug: placebo
- ICS/LABA FDC Dosage 2 (Active Comparator): High dose
  Interventions: Drug: placebo; Drug: fluticasone propionate; Drug: salmeterol

INTERVENTIONS:
Drug: fluticasone propionate — low dose
  Arms: ICS/LABA FDC Dosage 1
Drug: salmeterol
  Arms: ICS/LABA FDC Dosage 1
Drug: placebo — placebo/dummy for blinding purposes
  Arms: T+O FDC dosage 2
Drug: placebo — placebo/dummy for blinding purposes
  Arms: ICS/LABA FDC Dosage 2
Drug: tiotropium — tiotropium high dose
  Arms: T+O FDC dosage 2
Drug: olodaterol
  Arms: T+O FDC dosage 1
Drug: olodaterol
  Arms: T+O FDC dosage 2
Drug: placebo — placebo/dummy for blinding purposes
  Arms: T+O FDC dosage 1
Drug: placebo — placebo/dummy for blinding purposes
  Arms: ICS/LABA FDC Dosage 1
Drug: tiotropium — tiotropium low dose
  Arms: T+O FDC dosage 1
Drug: fluticasone propionate — low dose
  Arms: ICS/LABA FDC Dosage 2
Drug: salmeterol
  Arms: ICS/LABA FDC Dosage 2

SUMMARY:
The objective of the trial is to compare the lung function profile of once daily treatment with tiotropium+olodaterol FDC [2.5/ 5µg and 5/ 5µg] delivered by the RESPIMAT with the lung function profile of twice daily treatment with fluticasone propionate+salmeterol FDC [250/50µg and 500/50µg] delivered by the Accuhaler® after 6 weeks of treatment.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of chronic obstructive pulmonary disease
2. Relatively stable airway obstruction with a post-bronchodilator 30% </= Forced Expiratory Volume in 1 second (FEV1)<80% of predicted normal and a post-bronchodilator FEV1/(Forced Vital Capacity)FVC <70%
3. Male or female patients, 40 years of age or older
4. Smoking history of more than 10 pack years
5. Ability to perform technically acceptable pulmonary function tests and maintain records
6. Ability to inhale medication in a competent manner from the RESPIMAT Inhaler, Accuhaler and from a metered dose inhaler (MDI)

Exclusion criteria:

1. Significant disease other than COPD
2. COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or iv) or hospitalization in the last 3 months.
3. Clinically relevant abnormal lab values
4. History of asthma
5. Diagnosis of thyrotoxicosis
6. Diagnosis of paroxysmal tachycardia
7. History of myocardial infarction
8. Unstable or life-threatening cardiac arrhythmia
9. Hospitalization for heart failure within the past year
10. Known active tuberculosis
11. malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years
12. History of life-threatening pulmonary obstruction
13. History of cystic fibrosis
14. Clinically evident bronchiectasis
15. History of significant alcohol or drug abuse
16. History of thoracotomy with pulmonary resection
17. oral or patch ß-adrenergics
18. Oral corticosteroid medication within 6 weeks prior to Visit 1
19. Regular use daytime oxygen therapy for more than one hour per day
20. Pulmonary rehabilitation program in the six weeks prior to the screening visit
21. Investigational drug within one month or six half lives (whichever is greater) prior to screening visit
22. Known hypersensitivity to ß-adrenergic drugs, BAC, EDTA
23. Pregnant or nursing women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (29):
- Belgium (2):
  - 1237.11.32002 Boehringer Ingelheim Investigational Site, Genk
  - 1237.11.32001 Boehringer Ingelheim Investigational Site, Ghent
- Czechia (4):
  - 1237.11.42003 Boehringer Ingelheim Investigational Site, Kyjov
  - 1237.11.42004 Boehringer Ingelheim Investigational Site, Rokycany
  - 1237.11.42002 Boehringer Ingelheim Investigational Site, Tábor
  - 1237.11.42001 Boehringer Ingelheim Investigational Site, Třebíč
- Denmark (4):
  - 1237.11.45002 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1237.11.45004 Boehringer Ingelheim Investigational Site, Kolding
  - 1237.11.45001 Boehringer Ingelheim Investigational Site, Odense C
  - 1237.11.45003 Boehringer Ingelheim Investigational Site, Silkeborg
- Germany (5):
  - 1237.11.49003 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1237.11.49005 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.11.49001 Boehringer Ingelheim Investigational Site, Mannheim
  - 1237.11.49004 Boehringer Ingelheim Investigational Site, Mönchengladbach
  - 1237.11.49002 Boehringer Ingelheim Investigational Site, Wiesbaden
- Hungary (4):
  - 1237.11.36001 Boehringer Ingelheim Investigational Site, Debrecen
  - 1237.11.36004 Boehringer Ingelheim Investigational Site, Pécs
  - 1237.11.36003 Boehringer Ingelheim Investigational Site, Szeged
  - 1237.11.36002 Boehringer Ingelheim Investigational Site, Szombathely
- Netherlands (6):
  - 1237.11.31005 Boehringer Ingelheim Investigational Site, Almelo
  - 1237.11.31002 Boehringer Ingelheim Investigational Site, Breda
  - 1237.11.31006 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1237.11.31001 Boehringer Ingelheim Investigational Site, Heerlen
  - 1237.11.31007 Boehringer Ingelheim Investigational Site, Hoorn
  - 1237.11.31003 Boehringer Ingelheim Investigational Site, Zutphen
- Spain (3):
  - 1237.11.34003 Boehringer Ingelheim Investigational Site, Alicante
  - 1237.11.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1237.11.34002 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
- 1237.11.46001 Boehringer Ingelheim Investigational Site, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, double-dummy, active-controlled, 4-treatment, 4-period, complete cross-over design.
Pre-assignment Details: After signing informed consent, patients entered a 4-week screening period to ensure clinical stability (i.e. no exacerbations).
Groups:
- T+O 2.5/5 / T+O 5/5 / F+S 250/50 / F+S 500/50: Patients received a total of four treatments. Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days. The treatments were orally inhaled .
  * Fixed Dose Combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo (T+O 2.5/5).
  * Fixed dose combination (FDC) of Tiotropium 5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo (T+O 5/5).
  * Fixed dose combination (FDC) of Fluticasone propionate 250 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo (F+S 250/50).
  * Fixed dose combination (FDC) of Fluticasone propionate 500 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo (F+S 500/50).
  Tiotropium+Olodaterol FDC inhalation solutions were administered via the Respimat® inhaler once daily, Fluticasone propionate+Salmeterol FDC inhalation powders were administered orally twice daily via Accuhaler®.
- T+O 5/5 / F+S 500/50 / T+O 2.5/5 / F+S 250/50: Patients received a total of four treatments. Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days. The treatments were orally inhaled.
  * Fixed dose combination (FDC) of Tiotropium 5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo.
  * Fixed dose combination (FDC) of Fluticasone propionate 500 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo.
  * Fixed Dose Combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo.
  * Fixed dose combination (FDC) of Fluticasone propionate 250 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo.
  Tiotropium+Olodaterol FDC inhalation solutions were administered via the Respimat® inhaler once daily, Fluticasone propionate+Salmeterol FDC inhalation powders were administered orally twice daily via Accuhaler®.
- F+S 250/50 / T+O 2.5/5 / F+S 500/50 / T+O 5/5: Patients received a total of four treatments. Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days. The treatments were orally inhaled.
  * Fixed dose combination (FDC) of Fluticasone propionate 250 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo.
  * Fixed Dose Combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo.
  * Fixed dose combination (FDC) of Fluticasone propionate 500 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo.
  * Fixed dose combination (FDC) of Tiotropium 5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo.
  Tiotropium+Olodaterol FDC inhalation solutions were administered via the Respimat® inhaler once daily, Fluticasone propionate+Salmeterol FDC inhalation powders were administered orally twice daily via Accuhaler®.
- F+S 500/50 / F+S 250/50 / T+O 5/5 / T+O 2.5/5: Patients received a total of four treatments. Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days. The treatments were orally inhaled.
  * Fixed dose combination (FDC) of Fluticasone propionate 500 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo.
  * Fixed dose combination (FDC) of Fluticasone propionate 250 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo.
  * Fixed dose combination (FDC) of Tiotropium 5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo.
  * Fixed Dose Combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo.
  Tiotropium+Olodaterol FDC inhalation solutions were administered via the Respimat® inhaler once daily, Fluticasone propionate+Salmeterol FDC inhalation powders were administered orally twice daily via Accuhaler®.
Period: Overall Study
Arm/Group | T+O 2.5/5 / T+O 5/5 / F+S 250/50 / F+S 500/50 | T+O 5/5 / F+S 500/50 / T+O 2.5/5 / F+S 250/50 | F+S 250/50 / T+O 2.5/5 / F+S 500/50 / T+O 5/5 | F+S 500/50 / F+S 250/50 / T+O 5/5 / T+O 2.5/5
Started | 58 | 69 | 50 | 52
Completed | 54 | 57 | 45 | 46
Not Completed | 4 | 12 | 5 | 6
Not completed — Adverse Event | 3 | 8 | 3 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Non compliant with protocol | 1 | 1 | 0 | 2
Not completed — Other not defined above | 0 | 2 | 0 | 0
Not completed — Discontinued during washout periods. | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Treated Set: All randomised patients who received any dose of the trial medication.
Groups:
- Overall Study: Patients received a total of four treatments. Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days. The treatments were orally inhaled.
  * Fixed Dose Combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo.
  * Fixed dose combination (FDC) of Tiotropium 5 μg and Olodaterol 5 μg plus Fluticasone propionate+Salmeterol placebo.
  * Fixed dose combination (FDC) of Fluticasone propionate 250 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo.
  * Fixed dose combination (FDC) of Fluticasone propionate 500 μg and Salmeterol 50 μg plus Tiotropium+Olodaterol placebo.
  Tiotropium+Olodaterol FDC inhalation solutions were administered via the Respimat® inhaler once daily, Fluticasone propionate+Salmeterol FDC inhalation powders were administered orally twice daily via Accuhaler®.
Arm/Group | Overall Study
Number analyzed (Participants) | 229
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 148

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC (0-12h) Change From Patient Baseline After 6 Weeks of Treatment
Description: Change from patient baseline in Forced Expiratory Volume in one second (FEV1) Area Under the FEV1-time Curve from 0 to 12hours post-dose (AUC 0-12h) [L] after 6 weeks of treatment. Measured values presented are actually adjusted means.
  The period baseline is defined as the pre-dose measurement taken at on the day 1 of each period. The patient baseline is defined as the mean of non-missing period baselines for each patient.
Time Frame: Baseline and 6 weeks.
Population: FAS (Full Analysis Set): Included all randomised patients who were documented to have had received any dose of trial medication and who had both baseline and any evaluable post-baseline measurement for the primary efficacy endpoint.
Measure: Mean (Standard Error); unit: Litres
Groups:
- T+O 2.5/5 / F+S Placebo: Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days.
  • Fixed Dose Combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg (T+O 2.5/5) administered orally via the Respimat® inhaler once daily plus Fluticasone propionate+Salmeterol (F+S) placebo treatment administered orally twice daily via Accuhaler®.
- T+O 5/5 / F+S Placebo: Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days.
  • Fixed dose combination (FDC) of Tiotropium 5 μg and Olodaterol 5 μg (T+O 5/5) administered orally via the Respimat® inhaler once daily plus Fluticasone propionate+Salmeterol (F+S) placebo treatment administered orally twice daily via Accuhaler®.
- F+S 250/50 / T+O Placebo: Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days.
  • Fixed dose combination (FDC) of Fluticasone propionate 250 μg and Salmeterol 50 μg (F+S 250/50) administered orally twice daily via Accuhaler® plus Tiotropium+Olodaterol (T+O) placebo treatment administered orally once daily via the Respimat® inhaler.
- F+S 500/50 / T+O Placebo: Treatments were taken for 6 weeks and each treatment period was separated by a washout period of at least 21 days.
  • Fixed dose combination (FDC) of Fluticasone propionate 500 μg and Salmeterol 50 μg (F+S 500/50) administered orally twice daily via Accuhaler® plus Tiotropium+Olodaterol (T+O) placebo treatment administered orally once daily via the Respimat® inhaler.
Arm/Group | T+O 2.5/5 / F+S Placebo | T+O 5/5 / F+S Placebo | F+S 250/50 / T+O Placebo | F+S 500/50 / T+O Placebo
Number analyzed (Participants) | 214 | 216 | 211 | 217
Litres | 0.295 (0.014) | 0.317 (0.014) | 0.192 (0.015) | 0.188 (0.014)
Statistical Analysis 1: Comparison: T+O 5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 0-12h change from patient baseline (Tiotropium + Olodaterol 5/5 µg) = Mean FEV1 AUC 0-12h change from patient baseline (Fluticasone propionate + Salmeterol 250/50 µg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is two-sided alpha=0.05; Compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom; Mean Difference (Net) = 0.125, 95% CI 2-sided [0.103 to 0.147], Standard Error of Mean 0.011 — Difference calculated as T+O 5/5 - F+S 250/50 adjusted mean FEV1 AUC 0-12h change from patient baseline (L)
Statistical Analysis 2: Comparison: T+O 5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 0-12h change from patient baseline (Tiotropium + Olodaterol 5/5 µg) = Mean FEV1 AUC 0-12h change from patient baseline (Fluticasone propionate + Salmeterol 500/50 µg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.129, 95% CI 2-sided [0.107 to 0.150], Standard Error of Mean 0.011 — Difference calculated as T+O 5/5 - F+S 500/50 adjusted mean FEV1 AUC 0-12h change from patient baseline (L)
Statistical Analysis 3: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 0-12h change from patient baseline (Tiotropium + Olodaterol 2.5/5 µg) = Mean FEV1 AUC 0-12h change from patient baseline (Fluticasone propionate + Salmeterol 250/50 µg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.103, 95% CI [0.081 to 0.124], Standard Error of Mean 0.011 — Difference calculated as T+O 2.5/5 - F+S 250/50 adjusted mean FEV1 AUC 0-12h change from patient baseline (L)
Statistical Analysis 4: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 0-12h change from patient baseline (Tiotropium + Olodaterol 2.5/5 µg) = Mean FEV1 AUC 0-12h change from patient baseline (Fluticasone propionate + Salmeterol 500/50 µg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.106, 95% CI 2-sided [0.085 to 0.128], Standard Error of Mean 0.011 — Difference calculated as T+O 2.5/5 - F+S 500/50 adjusted mean FEV1 AUC 0-12h change from patient baseline (L)

2. Secondary Outcome: FEV1 AUC (0-24h) Change From Patient Baseline After 6 Weeks of Treatment
Description: Change from patient baseline in Forced Expiratory Volume in one second (FEV1) Area Under the FEV1-time Curve from 0 to 24 hours post-dose (AUC 0-24h) [L] after 6 weeks of treatment.
  Measured values presented are actually adjusted means. The period baseline is defined as the pre-dose measurement taken at on the day 1 of each period. The patient baseline is defined as the mean of non-missing period baselines for each patient.
Time Frame: Baseline and 6 weeks.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litres
Arm/Group | T+O 2.5/5 / F+S Placebo | T+O 5/5 / F+S Placebo | F+S 250/50 / T+O Placebo | F+S 500/50 / T+O Placebo
Number analyzed (Participants) | 214 | 216 | 211 | 217
Litres | 0.228 (0.014) | 0.244 (0.014) | 0.162 (0.014) | 0.159 (0.014)
Statistical Analysis 1: Comparison: T+O 5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 0-24h change from patient baseline (Tiotropium + Olodaterol 5/5 μg) = Mean FEV1 AUC 0-24h change from patient baseline (Fluticasone propionate + Salmeterol 250/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = 0.082, 95% CI 2-sided [0.061 to 0.103], Standard Error of Mean 0.011 — Difference calculated as T+O 5/5 - F+S 250/50 adjusted mean FEV1 AUC 0-24h change from patient baseline (L)
Statistical Analysis 2: Comparison: T+O 5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 0-24h change from patient baseline (Tiotropium + Olodaterol 5/5 μg) = Mean FEV1 AUC 0-24h change from patient baseline (Fluticasone propionate + Salmeterol 500/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.086, 95% CI 2-sided [0.065 to 0.107], Standard Error of Mean 0.011 — Difference calculated as T+O 5/5 - F+S 500/50 adjusted mean FEV1 AUC 0-24h change from patient baseline (L)
Statistical Analysis 3: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 0-24h change from patient baseline (Tiotropium + Olodaterol 2.5/5 μg) = Mean FEV1 AUC 0-24h change from patient baseline (Fluticasone propionate + Salmeterol 250/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.065, 95% CI 2-sided [0.045 to 0.086], Standard Error of Mean 0.011 — Difference calculated as T+O 2.5/5 - F+S 250/50 adjusted mean FEV1 AUC 0-24h change from patient baseline (L)
Statistical Analysis 4: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 0-24h change from patient baseline (Tiotropium + Olodaterol 2.5/5 μg) = Mean FEV1 AUC 0-24h change from patient baseline (Fluticasone propionate + Salmeterol 500/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.069, 95% CI 2-sided [0.048 to 0.090], Standard Error of Mean 0.011 — Difference calculated as T+O 2.5/5 - F+S 500/50 adjusted mean FEV1 AUC 0-24h change from patient baseline (L)

3. Secondary Outcome: Trough FEV1 Change From Patient Baseline After 6 Weeks of Treatment
Description: Change from patient baseline in Trough Forced Expiratory Volume in one second (FEV1) after 6 weeks of treatment. Trough FEV1 was defined as the mean of the 23h and 23h 50min (minutes) post-dose FEV1 measurements. Measured values presented are actually adjusted means.
  The period baseline is defined as the pre-dose measurement taken at on the day 1 of each period. The patient baseline is defined as the mean of non-missing period baselines for each patient.
Time Frame: Baseline and 6 weeks.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litres
Arm/Group | T+O 2.5/5 / F+S Placebo | T+O 5/5 / F+S Placebo | F+S 250/50 / T+O Placebo | F+S 500/50 / T+O Placebo
Number analyzed (Participants) | 214 | 216 | 211 | 217
Litres | 0.192 (0.014) | 0.197 (0.014) | 0.150 (0.014) | 0.139 (0.014)
Statistical Analysis 1: Comparison: T+O 5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean trough FEV1 change from patient baseline (Tiotropium + Olodaterol 5/5 μg) = Mean trough FEV1 change from patient baseline (Fluticasone propionate + Salmeterol 250/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.047, 95% CI 2-sided [0.022 to 0.071], Standard Error of Mean 0.012 — Difference calculated as T+O 5/5 - F+S 250/50 adjusted mean trough FEV1 change from patient baseline (L)
Statistical Analysis 2: Comparison: T+O 5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean trough FEV1 change from patient baseline (Tiotropium + Olodaterol 5/5 μg) = Mean trough FEV1 change from patient baseline (Fluticasone propionate + Salmeterol 500/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.058, 95% CI 2-sided [0.034 to 0.082], Standard Error of Mean 0.012 — Difference calculated as T+O 5/5 - F+S 500/50 adjusted mean trough FEV1 change from patient baseline (L)
Statistical Analysis 3: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean trough FEV1 change from patient baseline (Tiotropium + Olodaterol 2.5/5 μg) = Mean trough FEV1 change from patient baseline (Fluticasone propionate + Salmeterol 250/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.042, 95% CI 2-sided [0.018 to 0.067], Standard Error of Mean 0.012 — Difference calculated as T+O 2.5/5 - F+S 250/50 adjusted mean trough FEV1 change from patient baseline (L)
Statistical Analysis 4: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean trough FEV1 change from patient baseline (Tiotropium + Olodaterol 2.5/5 μg) = Mean trough FEV1 change from patient baseline (Fluticasone propionate + Salmeterol 500/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.054, 95% CI 2-sided [0.029 to 0.078], Standard Error of Mean 0.012 — Difference calculated as T+O 2.5/5 - F+S 500/50 adjusted mean trough FEV1 change from patient baseline (L)

4. Secondary Outcome: FEV1 AUC (12-24h) Change From Patient Baseline After 6 Weeks of Treatment
Description: Change from patient baseline in Forced Expiratory Volume in one second (FEV1) Area Under the FEV1-time Curve from 12 to 24 hours post-dose (AUC 12-24h) [L] after 6 weeks of treatment. Measured values presented are actually adjusted means.
  The period baseline is defined as the pre-dose measurement taken at on the day 1 of each period. The patient baseline is defined as the mean of non-missing period baselines for each patient.
Time Frame: Baseline and 6 weeks.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litres
Arm/Group | T+O 2.5/5 / F+S Placebo | T+O 5/5 / F+S Placebo | F+S 250/50 / T+O Placebo | F+S 500/50 / T+O Placebo
Number analyzed (Participants) | 214 | 216 | 211 | 217
Litres | 0.160 (0.014) | 0.172 (0.014) | 0.132 (0.014) | 0.129 (0.014)
Statistical Analysis 1: Comparison: T+O 5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 12-24h change from patient baseline (Tiotropium + Olodaterol 5/5 μg) = Mean FEV1 AUC 12-24h change from patient baseline (Fluticasone propionate + Salmeterol 250/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.039, 95% CI 2-sided [0.017 to 0.062], Standard Error of Mean 0.012 — Difference calculated T+O 5/5 - F+S 250/50 adjusted mean FEV1 AUC 12-24h change from patient baseline (L)
Statistical Analysis 2: Comparison: T+O 5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 12-24h change from patient baseline (Tiotropium + Olodaterol 5/5 μg) = Mean FEV1 AUC 12-24h change from patient baseline (Fluticasone propionate + Salmeterol 500/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.043, 95% CI 2-sided [0.021 to 0.065], Standard Error of Mean 0.011 — Difference calculated as T+O 5/5 - F+S 500/50 adjusted mean FEV1 AUC 12-24h change from patient baseline (L)
Statistical Analysis 3: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 12-24h change from patient baseline (Tiotropium + Olodaterol 2.5/5 μg) = Mean FEV1 AUC 12-24h change from patient baseline (Fluticasone propionate + Salmeterol 250/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p = 0.0146, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.028, 95% CI 2-sided [0.006 to 0.051], Standard Error of Mean 0.011 — Difference calculated as T+O 2.5/5 - F+S 250/50 adjusted mean FEV1 AUC 12-24h change from patient baseline (L)
Statistical Analysis 4: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean FEV1 AUC 12-24h change from patient baseline (Tiotropium + Olodaterol 2.5/5 μg) = Mean FEV1 AUC 12-24h change from patient baseline (Fluticasone propionate + Salmeterol 500/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p = 0.0055, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.032, 95% CI 2-sided [0.009 to 0.054], Standard Error of Mean 0.011 — Difference calculated as T+O 2.5/5 - F+S 500/50 adjusted mean FEV1 AUC 12-24h change from patient baseline (L)

5. Secondary Outcome: FEV1 Peak (0-3h) Change From Patient Baseline After 6 Weeks of Treatment
Description: Change from patient baseline in Forced Expiratory Volume in one second (FEV1) peak (0-3 hours) after 6 weeks of treatment. FEV1 peak (0-3 hours) was defined as the maximum FEV1 value measured within the first three hours post dosing. Measured values presented are actually adjusted means.
Time Frame: Baseline and 6 weeks.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litres
Arm/Group | T+O 2.5/5 / F+S Placebo | T+O 5/5 / F+S Placebo | F+S 250/50 / T+O Placebo | F+S 500/50 / T+O Placebo
Number analyzed (Participants) | 214 | 216 | 211 | 217
Litres | 0.401 (0.016) | 0.432 (0.016) | 0.291 (0.016) | 0.285 (0.015)
Statistical Analysis 1: Comparison: T+O 5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean FEV1 peak (0-3h) change from patient baseline (Tiotropium + Olodaterol 5/5 μg) = Mean FEV1 peak (0-3h) change from patient baseline (Fluticasone propionate + Salmeterol 250/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.142, 95% CI 2-sided [0.118 to 0.166], Standard Error of Mean 0.012 — Difference calculated as T+O 5/5 - F+S 250/50 adjusted mean FEV1 peak (0-3h) change from patient baseline (L)
Statistical Analysis 2: Comparison: T+O 5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean FEV1 peak (0-3h) change from patient baseline (Tiotropium + Olodaterol 5/5 μg) = Mean FEV1 peak (0-3h) change from patient baseline (Fluticasone propionate + Salmeterol 500/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.147, 95% CI 2-sided [0.123 to 0.171], Standard Error of Mean 0.012 — Difference calculated as T+O 5/5 - F+S 500/50 adjusted mean FEV1 peak (0-3h) change from patient baseline (L)
Statistical Analysis 3: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 250/50 / T+O Placebo; Null hypothesis: Mean FEV1 peak (0-3h) change from patient baseline (Tiotropium + Olodaterol 2.5/5 μg) = Mean FEV1 peak (0-3h) change from patient baseline (Fluticasone propionate + Salmeterol 250/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.111, 95% CI 2-sided [0.087 to 0.135], Standard Error of Mean 0.012 — Difference calculated as T+O 2.5/5 - F+S 250/50 adjusted mean FEV1 peak (0-3h) change from patient baseline (L)
Statistical Analysis 4: Comparison: T+O 2.5/5 / F+S Placebo vs F+S 500/50 / T+O Placebo; Null hypothesis: Mean FEV1 peak (0-3h) change from patient baseline (Tiotropium + Olodaterol 2.5/5 μg) = Mean FEV1 peak (0-3h) change from patient baseline (Fluticasone propionate + Salmeterol 500/50 μg). Hypothesis was analysed using a restricted maximum likelihood-based mixed effect repeated measures model including fixed effects of treatment and period; period baseline and patient baseline as covariates; patient as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.116, 95% CI 2-sided [0.092 to 0.140], Standard Error of Mean 0.012 — Difference calculated as T+O 2.5/5 - F+S 500/50 adjusted mean FEV1 peak (0-3h) change from patient baseline (L)

ADVERSE EVENTS:
Time Frame: From first drug intake until 21 days after last drug intake, up to 88 days.
Description: AEs are displayed by treatment, however in total patients were in the study for up to 223 days
Arm/Group | T+O 2.5/5 / F+S Placebo | T+O 5/5 / F+S Placebo | F+S 250/50 / T+O Placebo | F+S 500/50 / T+O Placebo
Serious Adverse Events (participants affected / at risk) | 6/215 | 7/221 | 4/212 | 9/219
Other Adverse Events (participants affected / at risk) | 21/215 | 28/221 | 19/212 | 24/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T+O 2.5/5 / F+S Placebo (N=215) | T+O 5/5 / F+S Placebo (N=221) | F+S 250/50 / T+O Placebo (N=212) | F+S 500/50 / T+O Placebo (N=219)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T+O 2.5/5 / F+S Placebo (N=215) | T+O 5/5 / F+S Placebo (N=221) | F+S 250/50 / T+O Placebo (N=212) | F+S 500/50 / T+O Placebo (N=219)
Nasopharyngitis (Infections and infestations) | 12 | 12 | 13 | 11
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 7 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.